CLINICAL TRIAL: NCT01430858
Title: Measurement of Induced Strains in the Human Tibia During Vibration Therapy and Habitual Activities
Brief Title: Does Vibration Therapy Induce Higher Than Normal Bone Strains and Strain Rates Than Those Experienced During Habitual Daily Activities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STH15516
Record Dates: First submitted 2011-09-07; First posted 2011-09-08 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Osteoporosis
Keywords: Fracture; Anabolic; Vibration; Strain Gauge; Focus - Osteoporosis
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Strain Gauge (Other): We wish to determine the relationship between tibial bone strain (recorded from implanted tibial strain gauges) and measured displacements of the limb and pelvis (using video motion analysis) during vibration exercise and a range of habitual locomotor activities. Only healthy volunteers will be recruited to this one arm.
  Interventions: Device: Strain Gauge; Other: Vibration therapy

INTERVENTIONS:
Device: Strain Gauge — The study participants will each undergo sterile surgical implantation of a tibial bone strain gauge in the right leg (dominance will recorded and determined by handedness). A single stacked, 45°, rosette strain gauge (FRA-2-11 Tokyo Sokki Kenkyujo Co., Japan) will be unilaterally bonded to the medial tibial cortex and carefully aligned with the long axis of the tibia. The gauge will be attached at the mid-shaft region, to determine the transmission of the vibrations through the bone and quantification of the microstructural effect.
  Other Names: Rosette strain gauge (FRA-2-11 Tokyo Sokki Kenkyujo Co., Japan)
Other: Vibration therapy — Galileo 900 platform. Study subjects will be asked to stand on the device for a series of 36 tests, with vibrations applied at various frequencies and amplitudes. A 20-second duration of videomotion & strain gauge readings will be captured.
  Juvent 1000 platform The volunteers will stand on the platform for one minute during which a 20-second duration of videomotion & strain gauge readings will be captured.
  Power Plate Pro5 Two amplitude settings will be tested, described as low & high. The subject will stand on each platform test for up to 1 minute, during which a 20-second duration of videomotion & strain gauge readings will be captured.
  Other Names: Galileo 900 platform (Novotec Medical GmbH, Medical device CE0123); Juvent 1000 platform (CE-marked); Power Plate Pro5 (CE-marked)

SUMMARY:
The overall aim of this study is to test the hypothesis that vibration exercise can induce higher than normal bone strains and strain rates than are experienced during habitual locomotor activities.

The investigators plan to study healthy young volunteers to:

1. Determine the relationship between tibial bone strain and

   * the frequency and amplitude of vibration therapy
   * a range of habitual locomotor activities;
2. Determine the transmission of vibrations during vibration therapy, in terms of

   * amplitude attenuation and phase shift of positional coordinates and accelerations at anatomic landmarks along the lower leg and other skeletal sites
   * the relationship between these and different frequencies and amplitudes of vibration therapy;
3. Determine the muscle power in the lower limb associated with various habitual locomotor activities and its relationship to the measured tibial bone strain.

The investigators subsequently hope to use the data captured in this experiment to develop a QCT-based finite element (FE) model of the human lower limb (tibia, fibula and foot). The investigators will then validate this model in relation to the characteristics (amplitude and phase shift) of the measured tibial bone strain and transmission of vibrations to the different anatomical landmarks during vibration therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, ages 18 to 50 years
* Generally healthy, as determined by review of medical history and physical exam
* Ambulatory
* Willing and physically able to undergo all study procedures
* BMD (measured by DXA) at the lumbar spine and hip within ± 2 SD of the young normal range
* BMI < 30

Exclusion Criteria:

* Previous diagnosis of osteoporosis
* History of fracture of the spine, pelvis, leg or foot
* History of bone or joint disorders affecting the shoulders, spine, pelvis, legs or feet (e.g. arthritis, congenital hip dislocation, spinal spondylolisthesis)
* Ongoing conditions or diseases known to cause secondary osteoporosis
* Malabsorption syndromes (e.g. coeliac or Crohn's disease)
* Known disorders of calcium metabolism
* Known history of thyroid disease
* Osteomalacia
* Paget's disease
* Diabetes
* History of cancer within the previous 5 years
* Epilepsy
* Ongoing conditions or use of medications that may impair vision or balance
* Use of the following medications within the previous 2 years

  * Bisphosphonates
  * Fluoride (except use for oral hygiene)
  * Strontium
  * Teriparatide
  * Other bone agents (e.g. SERMs, isoflavones, HRT, calcitonin etc)
  * Steroids
* Alcohol abuse or illicit drug use
* Pregnancy or currently trying to conceive (women only)
* Inability to give informed consent
* Known hypersensitivity to the antibiotic penicillin or cephalosporins
* Known hypersensitivity to the local anaesthetic lignocaine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum amplitudes of the vibrating principal strain, and maximum shear strain, γv (microstrain) of the tibial bone calculated from the tibial bone strains recorded during vibration therapy | At time of Vibration Therapy
Maximum principal strain εh and maximum shear strain γh (microstrain) of the tibial bone calculated from the tibial bone strains recorded during habitual locomotor activities | At time of Vibration Therapy

SECONDARY OUTCOMES:
Peak amplitude attenuation αv (in cm and percentage) and phase shift βv (in degrees) of the tibial strain primary endpoints εv and γv as a function of vibration frequency and amplitude (using the vibration device as a reference) | At time of Vibration Therapy
Peak amplitude attenuation and phase shift of the oscillating positional coordinates and accelerations | At time of Vibration Therapy
  Peak amplitude attenuation αm (in cm and percentage) and phase shift βm (in degrees) of the oscillating positional coordinates and accelerations (at different anatomical landmarks) measured by VICON MX motion analysis system during vibration therapy (using the vibration device as a reference)
Posture during vibration therapy assessed in terms of the angulations of the ankle, knee and hip joints and of the trunk, derived from the positional coordinates | At time of Vibration Therapy

CONTACTS AND LOCATIONS:
Overall Officials: Eugene McCloskey, Professor, Principal Investigator — University of Sheffield
Locations (1):
- Academic Unit of Bone Metabolism, Sheffield, South Yorks, United Kingdom